CLINICAL TRIAL: NCT04977219
Title: Prism Adaptation Training for Treatment of Spatial Neglect During Inpatient Rehabilitation
Status: Completed | Type: Observational
Sponsor: Sunnyview Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Robert Gillen, Clinical Neuropsychologist, Sunnyview Rehabilitation Hospital
Other Study IDs: 21-0505-3
Record Dates: First submitted 2021-07-09; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prism Adaptation Training;: Patients who received prism adaptation training for treatment of spatial neglect during their inpatient rehabilitation admission
  Interventions: Behavioral: Prism Adaptation Training
- Standard Care: Patients who received standard treatment of spatial neglect during their admission

INTERVENTIONS:
Behavioral: Prism Adaptation Training — Therapists administering PAT followed the protocol developed by the Kessler Foundation (2014).PAT sessions lasted approximately 30 minutes during which patients with left sided neglect don 20 diopter prism goggles deviating their visual field to the right while aiming their finger at a series of visual targets.
  Groups: Prism Adaptation Training;

SUMMARY:
Left sided spatial neglect is a common yet potentially debilitating phenomena associated with right hemisphere stroke. Heilman defines neglect as "the failure to report, respond, or orient to novel or meaningful stimuli presented to the side opposite of a brain lesion that cannot be attributed to either sensory or motor deficits". Numerous studies have demonstrated the impact of spatial neglect in right hemisphere stroke patients on both rehabilitation outcomes, and subsequent functioning in the community. Given the highly significant negative impact of spatial neglect, numerous treatment approaches have been attempted, yet most lack evidence in terms of efficacy. One promising exception has been prism adaptation training (PAT), which several recent reviews reported improved independence as a benefit of this treatment, both in terms of ameliorating the severity of neglect and demonstrating generalization to important functional behaviors. Still, much remains unknown regarding PAT, and not all studies have shown positive results.

At Sunnyview Rehabilitation Hospital, a number of providers have added PAT to the standard PT, OT and speech that stroke patients receive during their inpatient stay. As part of a process improvement initiative the investigators identified 57 patients that received PAT training between June 2016 and September of 2019. The investigators propose a retrospective case-control study examining the impact of PAT treatment on the rehabilitation outcomes for these patients. Outcome variables to be assessed include the measures of spatial neglect (Catherine Bergego Scale), functional independence measures (FIM), length of hospitalization and discharge destination. The investigators hypothesize that patients who received 4 or more PAT sessions during their inpatient rehabilitation stay will show improvements both in measures of neglect and functional independence as a result of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Right hemisphere stroke
* Admitted between 6/2016 & 12/2019

Exclusion Criteria:

* Absence of neglect
* Incomplete Catherine Bergego Scale (Less than 7 items scored)
* Evidence of traumatic brain injury
* Brain cancer
* Dementia
* Parkinson's disease
* Alzheimer's disease
* aphasia
* Interrupted hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient Rehabilitation Facility (IRF)
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Catherine Bergego Scale | Up to 55 days
  Behavioral measure of unilateral spatial neglect. Scored 0-30. Higher numbers indicate greater severity of spatial neglect.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Up to 55 days
  Measure of motoric and behavioral functioning of patients (eating, toileting, dressing, mobility). Scores range from 18-126. Higher scores indicate greater functional independence.
Length of Stay | Up to 55 days
  Length of inpatient hospital admission
Discharge destination | Up to 55 days
  Destination of patient following discharge: Home, Subacute nursing facility, Acute care hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillen RW, Harmon EY, Weil B, Fusco-Gessick B, Novak PP, Barrett AM. Prism Adaptation Treatment of Spatial Neglect: Feasibility During Inpatient Rehabilitation and Identification of Patients Most Likely to Benefit. Front Neurol. 2022 Apr 1;13:803312. doi: 10.3389/fneur.2022.803312. eCollection 2022. PMID 35432163